CLINICAL TRIAL: NCT03074383
Title: Improvement of Care for Outpatients With Type 2 Diabetes at the Porto Alegre Clinic Hospital Through Self-Care Multidisciplinary Workshop for Diabetes: a Randomized Controlled Trial
Brief Title: Improvement of Care for Outpatients With Type 2 Diabetes Through Self-Care Multidisciplinary Workshop for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0646
Record Dates: First submitted 2017-02-24; First posted 2017-03-08 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop (Experimental): Self-Care Multidisciplinary Workshop for Diabetes consist in individual meetings with a multidisciplinary team (nurse, pharmacist, nutritionist, physical educator, physiotherapist and social worker) in which education and self-care topics will be approached. The workshop will be offered in 3 different modules with 2-4 weeks difference between them.
  Interventions: Behavioral: Workshop
- Usual Care (Active Comparator): Usual care at outpatient Diabetes clinic AND 3 brief meetings with research team to receive printed educational material.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Workshop — A 15-minute Individual meetings with each professional (nurse, pharmacist, nutritionist, physical educator, physiotherapist and social worker) of the multidisciplinary team in which diabetes education and self-care topics will be approached.
  Other Names: Self-Care Multidisciplinary Workshop for Diabetes
  Arms: Workshop
Behavioral: Usual Care — Usual care at outpatient Diabetes clinic AND 3 brief meetings with research team to receive printed educational material.
  Arms: Usual Care

SUMMARY:
Ninety-six patients with diabetes will be randomly assigned to maintain standard treatment or participate in the Self-Care Multidisciplinary Workshop for Diabetes. The workshop consists of individual meetings, with a multidisciplinary team (nurse, pharmacist, nutritionist, physical educator and social worker) in which education and self-care topics will be approached aiming at the formation of knowledge and skills necessary for patient self-care. The workshop will be offered in 3 different modules with 2 to 4 weeks difference between them. The variation of glycated hemoglobin as well as aspects associated with self-care, adherence and quality of life will be evaluated at the study entry, 6 and 12 months later.

DETAILED DESCRIPTION:
Ninety-six patients with type 2 diabetes from our Diabetes Outpatient Clinic will be randomly assigned to maintain standard treatment or participate in the Self-Care Multidisciplinary Workshop for Diabetes. The workshop consists of 15-minute individual meetings with each professional of a multidisciplinary team (nurse, pharmacist, nutritionist, physical educator and social worker) in which education and self-care topics will be approached aiming at the formation of knowledge and skills necessary for patient self-care. The workshop will be offered in 3 different modules with 2 to 4 weeks difference between them.

Patients will be followed for 12 months. The variation of glycated hemoglobin as well as aspects associated with self-care, adherence and quality of life will be evaluated at the study entry, 6 and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous diagnosis of type 2 diabetes, HbA1c greater than 7.5% and age greater than 18 years

Exclusion Criteria:

* Types of diabetes other than type 2 diabetes; neurological, psychiatric or cognitive impairment that prevents proper understanding and participation in the workshop

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin from baseline at 12 months | 12 months
  Variation of glycated hemoglobin

SECONDARY OUTCOMES:
Change in glycated hemoglobin from baseline at 6 months | 6 months
  Variation of glycated hemoglobin
Variation of Diabetes Quality of Life Questionnaire from baseline at 6 months | 6 months
  Diabetes Quality of Life Questionnaire
Variation of Diabetes Quality of Life Questionnaire from baseline at 12 months | 12 months
  Diabetes Quality of Life Questionnaire
Glycated hemoglobin equal or less than 8,0 | 12 months
  Number of patients reaching glycated hemoglobin equal or less than 8,0
Glycated hemoglobin equal or less than 7,5 | 12 months
  Number of patients reaching glycated hemoglobin equal or less than 7,5
Variation of Summary of Diabetes Self-Care Activities Questionnaire (SDSCA) from baseline at 6 months | 6 months
  Change in SDSCA score 6 months after baseline
Variation of Summary of Diabetes Self-Care Activities Questionnaire (SDSCA) from baseline at 12 months | 12 months
  Change in SDSCA score 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz DAgord Schaan, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided